CLINICAL TRIAL: NCT03925077
Title: RERC on Technologies to Promote Exercise and Health Among People With Disabilities (A Scale Up Study Evaluating a Movement-to-Music Teleexercise Platform for Reaching a National Cohort of People With Spinal Cord Injury)
Brief Title: Spinal Cord Injury Program in Exercise
Acronym: SCIPE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Hui-Ju Young, PhD, Scientist, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: IRB-300003133; 90DPGE0005 (Other Grant/Funding Number: National Institute on Disability, Independent Living, and Rehabilitation Research)
Record Dates: First submitted 2019-03-27; First posted 2019-04-23 (Actual); Results first posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Spinal Cord Injuries
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded to participants' group assignments throughout the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Phase 1: Movement-to-Music (M2M) (Active Comparator): All M2M sessions are delivered using videos uploaded to a secure study website (the SCIPE website). Participants in M2M will have access to the website and attend three 60-minute M2M sessions per week for a total of 8 weeks. Each session provides rhythmic-based exercises that are choreographed to music to target range of motion, muscular strength, cardiorespiratory fitness, and balance. In addition, participants in M2M will receive and read weekly educational articles on health and fitness through the SCIPE website.
  Interventions: Other: Movement-to-Music
- Phase 1: Standard Exercise Training (SET) (Active Comparator): All SET sessions are delivered using videos uploaded to the SCIPE website. Participants in SET will have access to the website and attend three 60-minute SET sessions per week for a total of 8 weeks. Each session provides traditional exercises that target range of motion, muscular strength, cardiorespiratory fitness, and balance. In addition, participants in SET will receive and read weekly educational articles on health and fitness through the SCIPE website.
  Interventions: Other: Standard Exercise Training
- Phase 1: Attention Control (AC) (No Intervention): Participants in AC will not have access to any exercise videos. They will have access to the weekly educational articles on health and fitness, same as the ones received by the M2M and SET groups, through the SCIPE website.
- Phase 2: Standard Exercise Training (SET) (Active Comparator): All SET sessions are delivered using videos uploaded to the SCIPE website. Participants in SET will have access to the website and attend three 60-minute SET sessions per week for a total of 8 weeks. Each session provides traditional exercises that target range of motion, muscular strength, cardiorespiratory fitness, and balance. In addition, participants in SET will receive and read weekly educational articles on health and fitness through the SCIPE website.
  Interventions: Other: Standard Exercise Training
- Phase 2: Attention Control (AC) (No Intervention): Participants in AC will not have access to any exercise videos. They will have access to the weekly educational articles on health and fitness, same as the ones received by the M2M and SET groups, through the SCIPE website.

INTERVENTIONS:
Other: Movement-to-Music — The M2M program has been developed for onsite instruction and will be repurposed into an eHealth version. The program is based on the positive effects of exercise and music on both physiological and psychosocial outcomes in people with disabilities. Investigators aim to advance our current M2M program by enabling more robust personalization features, allowing people with SCI to individualize their M2M program. Movement and tempo-based adaptations will also be available. A typical M2M session will consist of tailored movement routines starting with a warmup using range of motion exercises, followed by muscle strengthening, cardiorespiratory, and/or balance routines, and ending with a cool down emphasizing breathing and mindfulness.
  Other Names: M2M
  Arms: Phase 1: Movement-to-Music (M2M)
Other: Standard Exercise Training — The SET program is based on the NCHPAD 14-Weeks to a Healthier You program launched in 2008. Exercise videos including range of motion, muscle strengthening, cardio and balance routines performed both seated and standing have been developed and will be restructured for use in this study. The SET program will be delivered through the same platform as M2M.
  Other Names: SET
  Arms: Phase 1: Standard Exercise Training (SET); Phase 2: Standard Exercise Training (SET)

SUMMARY:
The purpose of this study is to examine two 8-week, remotely delivered exercise interventions: Movement-to-Music (M2M) and Standard Exercise Training (SET), with 327 adults with spinal cord injury. Enrolled participants will be randomized into one of three groups: a) M2M, b) SET, and c) attention control (AC).

DETAILED DESCRIPTION:
The purpose of the Spinal Cord Injury Program in Exercise (SCIPE) study is to examine two 8-week, remotely delivered exercise interventions: Movement-to-Music (M2M) and Standard Exercise Training (SET), with 327 adults with SCI. The primary aim is to examine change in physical activity level after the 8-week M2M and SET interventions. We hypothesize that participants in M2M and SET will have significant increase in physical activity compared to an Attention Control (AC) group after the 8-week intervention. The secondary aim is to examine effects of the M2M and SET interventions on health and quality of life outcomes. We hypothesize that participants in M2M and SET will have significant increases in sleep quality and quality of life and decreases in pain and fatigue compared to AC after the 8-week intervention. Exercise enjoyment in M2M and SET participants will also be explored. The tertiary aim is to evaluate the demographic (age, race, sex), clinical (level of injury, type of injury), and psychosocial (social support, outcome expectations, self-efficacy, self-regulation) variables of two participant groups: 1) compliant participants who completed ≥ 50% of the intervention, and 2) noncompliant participants who completed post-testing but < 50% of the intervention or who did not complete post-testing.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed with a SCI resulting in incomplete or complete (C5 and below) paraplegia or tetraplegia;
2. Demonstrate readiness to physical activity by completing the Physical Activity Readiness Questionnaire for Everyone (PAR-Q+);
3. Obtain medical clearance if required by PAR-Q+;
4. Converse in and read English.

Exclusion Criteria:

1. No broadband internet access;
2. Significant visual impairment that prevents seeing a computer screen to follow a home exercise program;
3. Currently pregnant.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 96 (Actual)
Dates: Start 2021-02-01 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2025-03-31 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- RecTech Center, Birmingham, Alabama, United States

REFERENCES:
- [Derived] Young HJ, Mehta T, Kim Y, Padalabalanarayanan S, Chiu CY, Rimmer JH, Thirumalai M. The Spinal Cord Injury Program in Exercise (SCIPE) study: study protocol for a randomized controlled trial evaluating teleexercise programs for people with spinal cord injury. Trials. 2021 Aug 19;22(1):551. doi: 10.1186/s13063-021-05474-4. PMID 34412653

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited through social media platforms (e.g., Instagram, Facebook) and word of mouth. Recruitment for the Feasibility Phase took place between February 2021 and March 2022. Recruitment for the Effectiveness Phase occurred between August 2023 and September 2024. Recruitment and enrollment for both study phases were performed separately.
Pre-assignment Details: In the Feasibility Phase, the 36 enrolled participants were randomized to 3 groups: M2M, SET, and AC. For the Effectiveness Phase, the M2M arm was dropped after interim analysis and the 60 enrolled participants were randomized to 2 groups: SET and AC.
Period: Feasibility Phase
Arm/Group | Phase 1: Movement-to-Music (M2M) | Phase 1: Standard Exercise Training (SET) | Phase 1: Attention Control (AC) | Phase 2: Standard Exercise Training (SET) | Phase 2: Attention Control (AC)
Started | 12 | 12 | 12 | 0 | 0
8-week Assessment | 8 | 10 | 10 | 0 | 0
12-week Assessment | 5 | 8 | 9 | 0 | 0
16-week Assessment | 5 | 8 | 8 | 0 | 0
Completed | 5 | 8 | 8 | 0 | 0
Not Completed | 7 | 4 | 4 | 0 | 0
Not completed — Lost to Follow-up | 7 | 4 | 4 | 0 | 0
Period: Effectiveness Phase
Arm/Group | Phase 1: Movement-to-Music (M2M) | Phase 1: Standard Exercise Training (SET) | Phase 1: Attention Control (AC) | Phase 2: Standard Exercise Training (SET) | Phase 2: Attention Control (AC)
Started | 0 (In the Effectiveness Phase, the M2M was removed after discussing with the program officer. Hence, participants in the Effectiveness Phase were only randomized into either the SET arm or the AC arm.) | 0 (This cohort of participants was not part of the Feasibility Phase. The Effectiveness Phase recruited a new set of participants and performed a two-arm randomization (SET and AC).) | 0 (This cohort of participants was not part of the Feasibility Phase. The Effectiveness Phase recruited a new set of participants and performed a two-arm randomization (SET and AC).) | 30 | 30
8-week Assessment | 0 | 0 | 0 | 19 | 23
12-week Assessment | 0 | 0 | 0 | 22 | 22
16-week Assessment | 0 | 0 | 0 | 21 | 22
Completed | 0 | 0 | 0 | 21 | 22
Not Completed | 0 | 0 | 0 | 9 | 8
Not completed — Lost to Follow-up | 0 | 0 | 0 | 9 | 8

BASELINE CHARACTERISTICS:
Population: We report baseline characteristics of participants in the Effectiveness phase here. Approval was received from the program officer to remove the M2M arm from the Effectiveness phase, after completing the Feasibility phase with the 3 study arms (M2M, SET, and AC).
Groups:
- Phase 1: Movement-to-Music (M2M): All M2M sessions are delivered using videos uploaded to a secure study website (the SCIPE website). Participants in M2M will have access to the website and attend three 60-minute M2M sessions per week for a total of 8 weeks. Each session provides rhythmic-based exercises that are choreographed to music to target range of motion, muscular strength, cardiorespiratory fitness, and balance. In addition, participants in M2M will receive and read weekly educational articles on health and fitness through the SCIPE website.
  Movement-to-Music (M2M): The M2M program has been developed for onsite instruction and will be repurposed into an eHealth version. The program is based on the positive effects of exercise and music on both physiological and psychosocial outcomes in people with disabilities. Investigators aim to advance our current M2M program by enabling more robust personalization features, allowing people with SCI to individualize their M2M program. Movement and tempo-based adaptations will also be available. A typical M2M session will consist of tailored movement routines starting with a warmup using range of motion exercises, followed by muscle strengthening, cardiorespiratory, and/or balance routines, and ending with a cool down emphasizing breathing and mindfulness.
- Phase 1: Standard Exercise Training (SET): All SET sessions are delivered using videos uploaded to the SCIPE website. Participants in SET will have access to the website and attend three 60-minute SET sessions per week for a total of 8 weeks. Each session provides traditional exercises that target range of motion, muscular strength, cardiorespiratory fitness, and balance. In addition, participants in SET will receive and read weekly educational articles on health and fitness through the SCIPE website.
  Standard Exercise Training (SET): The SET program is based on the NCHPAD 14-Weeks to a Healthier You program launched in 2008. Exercise videos including range of motion, muscle strengthening, cardio and balance routines performed both seated and standing have been developed and will be restructured for use in this study. The SET program will be delivered through the same platform as M2M.
- Phase 2: Standard Exercise Training (SET): Standard Exercise Training (SET): The SET program is based on the NCHPAD 14-Weeks to a Healthier You program launched in 2008. Exercise videos including range of motion, muscle strengthening, cardio and balance routines performed both seated and standing have been developed and will be restructured for use in this study. The SET program will be delivered through the same platform as M2M.
- Total: Total of all reporting groups
Arm/Group | Phase 1: Movement-to-Music (M2M) | Phase 1: Standard Exercise Training (SET) | Phase 1: Attention Control (AC) | Phase 2: Standard Exercise Training (SET) | Phase 2: Attention Control (AC) | Total
Number analyzed (Participants) | 12 | 12 | 12 | 30 | 30 | 96
Age, Continuous [Mean (Standard Deviation); unit: Years] — Population: In Feasibility phase, there were three study arms (M2M, SET, and AC) with 36 participants randomized and participated. In the Effectiveness phase, the M2M arm was removed. The goal of the Effectiveness phase was to compare the effectiveness between SET and AC. We report the baseline characteristics of participants in the Effectiveness phase here.
  Years | 42.0 (11.6) | 47.7 (11.8) | 46.4 (12.0) | 49.5 (10.8) | 47.3 (12.3) | 47.3 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: In Feasibility phase, there were three study arms (M2M, SET, and AC) with 36 participants randomized and participated. In the Effectiveness phase, the M2M arm was removed. The goal of the Effectiveness phase was to compare the effectiveness between SET and AC. We report the baseline characteristics of participants in the Effectiveness phase here.
  Participants
    Female | 6 | 5 | 8 | 20 | 17 | 56
    Male | 6 | 7 | 4 | 10 | 13 | 40
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants] — Population: In Feasibility phase, there were three study arms (M2M, SET, and AC) with 36 participants randomized and participated. In the Effectiveness phase, the M2M arm was removed. The goal of the Effectiveness phase was to compare the effectiveness between SET and AC. We report the baseline characteristics of participants in the Effectiveness phase here.
  Participants
    Hispanic or Latino | 1 | 1 | 2 | 4 | 2 | 10
    Not Hispanic or Latino | 11 | 11 | 9 | 26 | 28 | 85
    Unknown or Not Reported | 0 | 0 | 1 | 0 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: In Feasibility phase, there were three study arms (M2M, SET, and AC) with 36 participants randomized and participated. In the Effectiveness phase, the M2M arm was removed. The goal of the Effectiveness phase was to compare the effectiveness between SET and AC. We report the baseline characteristics of participants in the Effectiveness phase here.
  Participants
    American Indian or Alaska Native | 0 | 0 | 2 | 0 | 0 | 2
    Asian | 1 | 0 | 0 | 0 | 1 | 2
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
    Black or African American | 1 | 2 | 2 | 7 | 6 | 18
    White | 10 | 10 | 6 | 20 | 22 | 68
    More than one race | 0 | 0 | 0 | 3 | 0 | 3
    Unknown or Not Reported | 0 | 0 | 2 | 0 | 1 | 3

OUTCOME MEASURES:

1. Primary Outcome: Physical Activity Level at Week 8
Description: Physical activity was assessed using the Leisure Time Physical Activity Questionnaire for People with Spinal Cord Injury (LTPAQ-SCI). The LTPAQ-SCI is a 3-item, self-report questionnaire that measures the minutes people with spinal cord injury spend in mild, moderate, and heavy intensity leisure time physical activity in the last 7 days.
Time Frame: Post 8-week intervention
Population: We report outcomes collected for the Effectiveness phase here. The goal of the Effectiveness phase was to compare the effectiveness between SET and AC. The M2M arm was removed per approval and participants enrolled in the Effectiveness phase were randomized to SET or AC.
Measure: Mean (Standard Deviation); unit: Minutes per week
Groups:
- Phase 2: Standard Exercise Training (SET): All M2M sessions are delivered using videos uploaded to the SCIPE website. Participants in SET will have access to the website and attend three 60-minute SET sessions per week for a total of 8 weeks. Each session provides traditional exercises that target range of motion, muscular strength, cardiorespiratory fitness, and balance. In addition, participants in M2M will receive and read weekly educational articles on health and fitness through the SCIPE website.
  Standard Exercise Training: The SET program is based on the NCHPAD 14-Weeks to a Healthier You program launched in 2008. Exercise videos including range of motion, muscle strengthening, cardio and balance routines performed both seated and standing have been developed and will be restructured for use in this study. The SET program will be delivered through the same platform as M2M.
Arm/Group | Phase 2: Standard Exercise Training (SET) | Phase 2: Attention Control (AC)
Number analyzed (Participants) | 20 | 21
Minutes per week | 383 (347) | 297 (227)

2. Secondary Outcome: Pain Intensity Week 8
Description: The pain intensity was assessed using the NIH Patient-Reported Outcomes Measurement Information System (PROMIS®) Pain Intensity Adult Short Form 3a (v1.0). The instrument is a 3-item measure with the response scores ranging from 1 (Had no pain) to 5 (Very severe). The total raw score is converted to a T-score (population mean=50, SD=10) using standard scoring guidelines for each participant for analysis. Higher scores indicate higher pain intensity.
Time Frame: Post 8-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 2: Standard Exercise Training (SET) | Phase 2: Attention Control (AC)
Number analyzed (Participants) | 20 | 23
T-score | 53.5 (10.6) | 56.3 (9.9)

3. Secondary Outcome: Pain Interference at Week 8
Description: The influence of pain on performing daily activities was assessed with the NIH Patient-Reported Outcomes Measurement Information System (PROMIS®) Pain Interference Adult Short Form 8a (v1.0). The form contains 8 items with 5 response options ranging from 1 (Not at all) to 5 (Very much). The form has raw scores range from 8 to 40, with higher scores indicating more pain interference. The total raw score is converted to a T-score (population mean=50, SD=10) using standard scoring guidelines for each participant for analysis.
Time Frame: Post 8-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 2: Standard Exercise Training (SET) | Phase 2: Attention Control (AC)
Number analyzed (Participants) | 20 | 23
T-score | 53.6 (8.5) | 55.5 (8.9)

4. Secondary Outcome: Sleep Quality at Week 8
Description: Sleep quality is assessed using the NIH Patient-Reported Outcomes Measurement Information System (PROMIS®) Sleep Disturbance Adult Short Form 8a, which contains 8 items on a 5-point Likert scale, ranging from 1 (Very much) to 5 (Not at all). The form has raw scores range from 8 to 40, with higher scores indicating worst sleep quality. The total raw score is converted to a T-score (population mean=50, SD=10) using standard scoring guidelines for each participant for analysis.
Time Frame: Post 8 week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 2: Standard Exercise Training (SET) | Phase 2: Attention Control (AC)
Number analyzed (Participants) | 20 | 23
T-score | 51.7 (5.6) | 52.7 (5.6)

5. Secondary Outcome: Fatigue Level at Week 8
Description: Fatigue was measured using the NIH Patient-Reported Outcomes Measurement Information System (PROMIS®) Fatigue Adult Short Form. The instrument is a 8 items on a 5-point Likert scale, ranging from 1 (Not at all/Never) to 5 (Very much/Always). Higher scores indicate higher fatigue. The total raw score is converted to a T-score (population mean=50, SD=10) using standard scoring guidelines for each participant for analysis.
Time Frame: Post 8-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 2: Standard Exercise Training (SET) | Phase 2: Attention Control (AC)
Number analyzed (Participants) | 20 | 23
T-score | 50.1 (10.5) | 55.1 (9.7)

6. Secondary Outcome: Health-related Physical Quality of Life at Week 8
Description: Health-related quality of life was assessed using the NIH Patient-Reported Outcomes Measurement Information System (PROMIS®) 10 Global Health Items. The Global-10 Health form is a 10-item measure with the response scores ranging from 1 (Poor/Not at all/Always/Very severe) to 5 (Excellent/Completely/Never/None). One question item, "how would you rate your pain on average?", is on a 11-point Likert scale that ranges from 0 (No pain) to 10 (Worst pain imaginable). Higher scores indicate better health-related quality of life. The total raw score is converted to a T-score (population mean=50, SD=10) using standard scoring guidelines for each participant for analysis.
Time Frame: Post 8-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 2: Standard Exercise Training (SET) | Phase 2: Attention Control (AC)
Number analyzed (Participants) | 20 | 23
T-score | 43.6 (8.5) | 41.3 (6.8)

7. Secondary Outcome: Ability to Participate in Social Roles and Activities at Week 8
Description: Social participation was measured using the NIH Patient-Reported Outcomes Measurement Information System (PROMIS®) Ability to Participate in Social Roles and Activities Short Form 8a. The instrument is a 8-item measure with the response scores ranging from 1 (always) to 5 (never). The lowest possible total raw score is 8 and the highest possible score is 40. Higher scores indicate better ability to participate in social roles and activities. The total raw score is converted to a T-score (population mean=50, SD=10) using standard scoring guidelines for each participant for analysis.each participant for analysis.
Time Frame: Post 8-week intervention
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Phase 2: Standard Exercise Training (SET) | Phase 2: Attention Control (AC)
Number analyzed (Participants) | 20 | 23
T-score | 50.3 (9.0) | 45.4 (9.4)

ADVERSE EVENTS:
Time Frame: From enrollment until end of week-16 follow up
Description: The SCIPE study monitored adverse events (AEs) and reported them based on four types defined by the Behavior Change Consortium of the National Institutes of Health. The four types of AEs are: 1) Falls; 2) Cardiovascular-related episodes; 3) Musculoskeletal-related events; and 4) Health care use. All AEs would be assessed for severity and causality and reported to IRB and relevant regulatory bodies when necessary.
Arm/Group | Phase 1: Movement-to-Music (M2M) | Phase 1: Standard Exercise Training (SET) | Phase 1: Attention Control (AC) | Phase 2: Standard Exercise Training (SET) | Phase 2: Attention Control (AC)
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/30 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/30 | 0/30
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12 | 0/12 | 0/30 | 0/30

LIMITATIONS AND CAVEATS:
Because the interventions were delivered asynchronously, it was challenging to verify whether participants consistently completed the exercises or engaged with the videos and articles. Maintaining long-term engagement after the intervention also proved challenging, highlighting the need for future research to identify factors contributing to attrition and to develop strategies that promote sustained participation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2023-07-22): https://cdn.clinicaltrials.gov/large-docs/77/NCT03925077/Prot_SAP_ICF_000.pdf